CLINICAL TRIAL: NCT01537692
Title: A Randomized, Open-Label, 3-Period Crossover Study to Investigate the Pharmacokinetics, Safety and Tolerability of BDP HFA Nasal Aerosol in Healthy Volunteers
Brief Title: Clinical Study to Evaluate the Pharmacokinetics and Safety of BDP HFA Nasal Aerosol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BDP-AR-101
Record Dates: First submitted 2012-02-15; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BDP HFA Nasal Aerosol 80 mcg/d (Experimental): single dose, intranasal aerosol
  Interventions: Drug: BDP HFA Nasal Aerosol
- BDP HFA Nasal Aerosol 320 mcg/d (Experimental): single dose, intranasal aerosol
  Interventions: Drug: BDP HFA Nasal Aerosol
- BDP HFA Inhalation Aerosol 320 mcg/d (Active Comparator): single dose, orally inhaled aerosol
  Interventions: Drug: BDP HFA Inhalation Aerosol (QVAR)

INTERVENTIONS:
Drug: BDP HFA Nasal Aerosol — BDP HFA Nasal 80mcg
  Arms: BDP HFA Nasal Aerosol 80 mcg/d
Drug: BDP HFA Nasal Aerosol — BDP HFA Nasal 320mcg
  Arms: BDP HFA Nasal Aerosol 320 mcg/d
Drug: BDP HFA Inhalation Aerosol (QVAR) — BDP HFA Oral 320mcg
  Arms: BDP HFA Inhalation Aerosol 320 mcg/d

SUMMARY:
The purpose of this study is to compare the systemic levels of beclomethasone 17 monopropionate (17 BMP - the active metabolite of BDP) after intranasal administration of BDP HFA with the systemic levels of 17 BMP after administration of orally inhaled BDP HFA in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Male or female subjects 18-45 years of age
* General good health

Exclusion Criteria:

* History of physical findings of nasal pathology (within 60 days prior to Screening Visit)
* Participation in any investigational drug study 30 days preceding Screening Visit
* History of respiratory infection/disorder with 28 days preceding Screening Visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 24 hours post dose
  * Area under the plasma concentration time curve until the last measurable value (AUClast) for 17-BMP
  * Maximum plasma concentration (Cmax) for 17-BMP

SECONDARY OUTCOMES:
Pharmacokinetics | 24 hours post dose
  * Area under the plasma concentration time curve extrapolated to infinity (AUC0-inf), time to mean peak plasma concentration (Tmax), and the terminal elimination half-life (t1/2) for 17-BMP
  * AUClast, AUC0-inf, Cmax, Tmax, t1/2 for BDP
Safety and tolerability of BDP HFA nasal aerosol | 24 hours post dose
  Change from baseline in safety and tolerability endpoints - including Adverse events, changes in vital signs (blood pressure and pulse rate) and ENT exams (every visit) and safety laboratory assessments and physical exams (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, PhD, Study Director — Teva Global Respiratory Research

REFERENCES:
- [Derived] Ratner PH, Melchior A, Dunbar SA, Tantry SK, Dorinsky PM. Pharmacokinetic profile of beclomethasone dipropionate hydrofluoroalkane after intranasal administration versus oral inhalation in healthy subjects: results of a single-dose, randomized, open-label, 3-period crossover study. Clin Ther. 2012 Jun;34(6):1422-31. doi: 10.1016/j.clinthera.2012.04.023. Epub 2012 May 22. PMID 22621776